CLINICAL TRIAL: NCT02142270
Title: Epidemiology of Sudden Cardiac Arrest in Sub-Saharan Africa: Rationale and Design
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cameroon Resuscitation Council (Other)
Responsible Party: Principal Investigator, BONNY Aimé, Principal investigator, Cameroon Resuscitation Council
Other Study IDs: PASCAR
Record Dates: First submitted 2014-05-10; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years

GROUPS / COHORTS (2):
- Victims of cardiac arrest, either SCD or aborted SCA
- Premature death: All residents of districts of interest will be surveyed during 3 years. premature deaths occurring in residents of districts of interest will be checked for past medical history, circumstances of death, and autopsy report (if possible). Investigators will also analyze the employment of resuscitation attempts during the timeframe of sudden cardiac arrest (SCA) in various patient populations throughout African countries.
  The arm group of the study is every resident of the district of interest

SUMMARY:
Background The burden of sudden cardiac death (SCD) in Africa is unknown. Our aim is to assess the epidemiology of SCD in Africa. Methods The sub-Saharan Africa SCD study is a prospective, multicenter, community-based registry monitoring all cases of cardiac arrest occurring in victims > 15 years old. Investigators will use the definition of established SCD if an unexpected death without obvious extracardiac cause, occurred with a rapid witnessed collapse, or if unwitnessed, occurred within 1 hour after the onset of symptoms; probable SCD if an unexpected death without obvious extracardiac cause occurred within the previous 24 hours. After approval from institutional boards, Investigators will record demographic, clinical, electrocardiographic and biological variables of SCD victims (including survivors of cardiac arrest) in several sub-Saharan African cities. All deaths occurring in residents of districts of interest will be checked for past medical history, circumstances of death, and autopsy report (if possible). Investigators will also analyze the employment of resuscitation attempts during the timeframe of sudden cardiac arrest (SCA) in various patient populations throughout countries. Conclusion This study will provide comprehensive, contemporary data on the epidemiology of SCD in sub-Saharan Africa and will help in the development of strategies to prevent and manage cardiac arrest in this region of the world.

ELIGIBILITY:
Inclusion Criteria:

* Victims of cardiac arrest, either SCD or aborted SCA

Exclusion Criteria:

* Age ≤ 15 years.
* Refusal of consent (by the family).

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All residents of districts of interest will be surveyed during 3 years. premature deaths occurring in residents of districts of interest will be checked for past medical history, circumstances of death, and autopsy report (if possible). Investigators will also analyze the employment of resuscitation attempts during the timeframe of sudden cardiac arrest (SCA) in various patient populations throughout African countries.
  The arm group of the study is every resident of the district of interest
Sampling Method: Non-Probability Sample
Enrollment: 250000 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Sudden Cardiac Death | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Bonny, Douala, Cameroon